CLINICAL TRIAL: NCT06052514
Title: Efficacy of CPAP in Reducing Cognitive Fog in Post-COVID Patients With Sleep Apnea
Brief Title: CPAP Efficacy in Post-COVID-19 Patients With Sleep Apnea
Acronym: BreathePA
Status: Completed | Type: Observational
Sponsor: Venkatesh Krishnamurthy (Other)
Collaborators: Breathe Pennsylvania (Unknown)
Responsible Party: Sponsor-Investigator, Venkatesh Krishnamurthy, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY23070113
Record Dates: First submitted 2023-09-21; First posted 2023-09-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Sleep Apnea
MeSH Terms: conditions — COVID-19; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Post COVID patient diagnosed with sleep apnea with AHI > 5: Patients with post COVID syndrome diagnosed with sleep apnea starting CPAP
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Patients with moderate or severe OSA will be treated with CPAP

SUMMARY:
This is a prospective, observational study evaluating the relationship between severity of sleep apnea with severity of cognitive fog and if treatment of sleep apnea with CPAP improves cognitive fog in a cohort of post COVID patients with sleep apnea.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to evaluate the extent to which OSA may be a common, treatable comorbidity in post-COVID patients suffering from cognitive fog and whether addressing the sleep apnea may help these patients in resolving this distressing symptom.

According to the World Health Organization (WHO), "post-COVID-19 condition occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset, with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis". It is estimated that up to 20 to 90% of post COVID patients will have at least one persisting symptom that lasts for more than 4 months. According to the WHO, the most common symptoms include, but are not limited to shortness of breath (78%), fatigue (78%), and cognitive dysfunction (74%). It has serious economic consequences as 46% of patients were working on a reduced schedule and 23% left the workforce. Though the underlying pathology is thought to be a pan-inflammatory response, the etiology can be multifactorial. OSA is one of the possible etiologies as its symptoms and underlying inflammatory pathophysiology overlaps with that of post COVID syndrome.

Obstructive sleep apnea (OSA), a pulmonary disorder in which patients have stopping breathing episodically at night, is common, occurring in up to 60% of post COVID 19 patients. Patients with preexisting OSA have a 59% and 89% chances of developing post COVID symptoms in men and women respectively. The intermittent 'stopping breathing' episodes, sleep fragmentation and intermittent hypoxia in patients with OSA triggers a persistent, chronic low-grade inflammation within the central nervous system leading to activation of microglia and astrocytes which in turn leads to synaptic loss, neuronal necrosis and apoptosis which manifests as cognitive deficits. Interestingly, post COVID syndrome presents with similar symptoms of difficulty breathing and cognitive fog, and is associated with a similar but independent, chronic inflammatory process in the central nervous system, leading to synaptic and neuronal loss and cognitive fog. When patients with pre-existing OSA have post COVID syndrome, there may be worsening of the cognitive fog because of synergistic increase in inflammatory responses. Further, treatment of sleep apnea with CPAP can improve cognitive fog as it could decrease the inflammatory response in post COVID patients with sleep apnea. Hence, it is important to understand the relationship between the severity of OSA to the severity of cognitive fog, and if CPAP treatment can decrease the cognitive fog, thereby improve quality of life in post COVID patients.

The investigator proposes to conduct a four-week longitudinal, observational pilot study in a sample of 30 patients with sleep apnea, recruited from the post COVID clinic over a period of one year. The investigator will evaluate the severity of cognitive fog at baseline and change in cognitive fog with CPAP treatment from baseline to four weeks of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years of age.
* Diagnosed with COVID and continues to have persistent symptoms beyond 4 weeks.
* Diagnosed with sleep apnea based on a home sleep study

Exclusion Criteria:

* Patients with Narcolepsy or other acute Primary sleep problems.
* Cognitive impairment secondary to a neurodegenerative disorders and dementia.
* Acute exacerbation of psychiatric illness including severe depression, schizophrenia or bipolar disorder in the past 30 days.
* Serious medical or neurological illness or infection requiring hospitalization or unable to function in the past 30 days.
* Any medications that were started or change in dosage of the following medication in the past 30 days including: corticosteroids, stimulants, benzodiazepines/non benzodiazepine receptor agonists, antidepressants, antipsychotics or other medications which alter cognition.
* Patients who are on any active treatment for sleep apnea including CPAP, dental device or implant for two weeks before enrolling into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the post COVID clinic run by the Comprehensive lung Clinic at the Falk building, University of Pittsburgh.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Montreal Cognitive Assessment at 4-6 Weeks | Baseline, 4-6 Weeks
  Cognitive Fog as measured on Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Change from Baseline Digit span backwards and sequential in at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring attention, concentration and working memory as measured on Digit span backwards and sequential
Change from Baseline in Trail making A and B test at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring selective and divided attention, working memory, visuospatial skills and psychomotor performance as measured on Trail making A and B test
Change from Baseline in Digit symbol substitution at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring intelligence, response speed, sustained attention, visual spatial skills and set shifting as measured on Digit symbol substitution
Change from Baseline in Benson complex figure at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring visuospatial abilities, visual memory and executive abilities as measured on Benson complex figure
Change from Baseline in Stroop color word test at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring executive functions of selective and focused attention, cognitive flexibility and inhibition as measured on Stroop color word test
Change from Baseline the psychomotor vigilance task (PVT) at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring alertness, problem solving and psychomotor skills as measured on the psychomotor vigilance task (PVT)
Change from Baseline Multilingual naming test (MINT) test at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring naming impairment as measured on the Multilingual naming test (MINT)
Change from Baseline Verbal fluency at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring speeded word retrieval to phonemic cues as measured on Verbal fluency
Change from Baseline Categorical fluency at 4-6 Weeks | Baseline, 4-6 Weeks
  Neuropsychological assessment measuring semantic memory as measured on Categorical fluency

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Krishnamurthy, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No